CLINICAL TRIAL: NCT04112615
Title: Project Aura: Co-design of a Home-based Monitoring Service for Patients With Chronic Kidney Disease
Brief Title: Project Aura: Co-design of a Home-based Monitoring Service
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 271364
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Anemia of Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients and/or carers: Patients and/or their nominated carers come in to give feedback on the device and the system as a whole, from usability to design.
  Interventions: Device: Blood measurement
- Healthcare professionals: Healthcare professionals come in to give feedback on the device and the system, from what results they would like to see and their concerns about patients using it.
  Interventions: Device: Blood measurement

INTERVENTIONS:
Device: Blood measurement — Single fingerprick to measure haemoglobin and haematocrit measurements using a potential haemoglobin home monitoring system.

SUMMARY:
Co-design of a home-based haemoglobin monitoring system with participants with anaemia of chronic kidney disease.

DETAILED DESCRIPTION:
The device/monitoring system being developed measures the haemoglobin and haematocrit levels in blood from a single drop of blood. By measuring these blood parameter, participants are able to monitor their haemoglobin level at home.

The use of the device will take place in the participant's home to simulate what the investigators believe will be the ideal location for people who would prefer to self-manage their condition.

This study is a unique opportunity to gain feedback on the future design and development of a home-based monitoring system through user evaluation. As this is an adaptive/ iterative study design, this will give the Sponsor the opportunity to make changes to the user interface and user platform based on the feedback received from the end user.

ELIGIBILITY:
Inclusion criteria:

For patients:

* Adequate English to participate in focus groups without an interpreter
* Patients of the study site who are currently undergoing treatment for anaemia of CKD
* Patients willing to participate in at least one or more 60-minute and ideally 90-minute focus groups at the designated study location, time and date.
* Patients capable of providing informed consent before attending the first focus group

For carers:

* Should be the primary carer nominated by a patient who fulfils the inclusion criteria, this includes parents of affected children
* Should be willing to participate in at least 60-minute and ideally 90-minute focus groups at the designated study location, time and date.
* Carers can only participate in the study with the patient he/she is caring for. The patient has also to be involved in the study
* Carers need to be capable of providing informed consent before attending the first focus group

For healthcare professionals:

* All clinicians need to be current employees of the study site
* Doctors need to be employed at Specialist Registrar, Fellow or Consultant Level
* Nurses of all grades are invited to participate but ideally need to have had some involvement in the outpatient care of CKD patients with anaemia

All participants:

* Should be willing to have the session's recorded audio, transcripts and analysed data from the focus groups shared with Entia.
* should be willing to attend multiple 60 to 90 minute focus groups.
* should be willing for unidentifiable photos and video footage to be taken during the interview.
* Participants attending focus groups later in the development process must be comfortable consenting to finger prick testing/ assessing the ease of use of the test disposable

Exclusion criteria:

Patients:

* Does not have adequate English to participate in focus group interviews without an interpreter.
* Patients of the study site who are not currently undergoing treatment or have previously undergone treatment within the past 12 months.
* Patients not willing to participate in at least 60-minute and ideally 90-minute focus group discussion at the designated study location, time and date.
* Participant not capable of providing consent or have a suitable, legally acceptable representative present to provide consent before the focus group interview.

For carers:

* Is not the nominated primary carer of a patient who fulfils the inclusion criteria, this includes parents of affected children
* Not paired with a patient that is involved in the study
* Carers not willing to participate in at least a 60-minute and ideally 90-minute focus group discussion at the designated study location, time and date.

For healthcare professionals:

None.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants will be recruited from the study site.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Qualitative capture of user feedback- focus groups | 12 months
  User feedback gathered from participants using the blood measurement device will be used to inform the changes necessary to develop a successful home-based haemoglobin monitoring system.
  Feedback will be analysed based on framework analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Bhandari, FHEA, Principal Investigator — Hull University Teaching Hospital
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only within clinical team involved in this study and design and research teams in Entia.